CLINICAL TRIAL: NCT00000342
Title: Risperidone for the Treatment of Cocaine Dependence
Brief Title: Risperidone for the Treatment of Cocaine Dependence - 7
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-3-0010-7; Y01-3-0010-7
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-16 (Estimated); Status verified 1997-06

CONDITIONS: Cocaine-Related Disorders
Keywords: cocaine dependence
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Risperidone

INTERVENTIONS:
Drug: Risperidone

SUMMARY:
The purpose of this study is to evaluate clinical safety and pharmacological efficacy in the treatment of cocaine dependence, to evaluate impact of treatment on craving, and to correlate evidence of baseline neurotoxic damage of cocaine with treatment outcome and clinical side-effects.

ELIGIBILITY:
Inclusion Criteria:

M/F ages 21-50. Meet DSM-IV criteria for cocaine dependence. Agree to conditions of the study and sign informed consent.

Exclusion Criteria:

Psychiatric disorder that requires medication therapy. History of seizures. Pregnant and/or nursing women. Dependence on ETOH or benzodiazepines or other sedative/hypnotics. Acute hepatitis. Other medical conditions that deem participation to be unsafe.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0
Dates: Start 1996-07; Primary Completion 1997-08 (Actual); Study Completion 1997-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Ling, M.D., Principal Investigator — Friends Research Institute, Inc.
Locations (1):
- Friends Research Institute, Los Angeles, California, United States